CLINICAL TRIAL: NCT05889286
Title: Phase II Investigation of [F-18]MHF as a PET Tracer to Detect Orthopedic Implants-associated Infection
Brief Title: F18-MHF: Orthopedic Implants-Associated Infection Detection
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mark M Goodman, Professor, Emory University
Other Study IDs: STUDY00006008; 5R42AI157552-03 (NIH)
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Knee Disease; Knee Infection
Keywords: Implant; Orthopedic implants; Implant Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm A: Symptomatic patient cohort: Arm A will consist of 20 patients who have suspected prosthetic infection and who are scheduled to undergo surgery debridement/removal.
  Interventions: Drug: [F-18]MHF
- Arm B: Asymptomatic patient cohort: Arm B will consist of 10 asymptomatic normal control patients who have remotely placed total knee prosthesis without clinical or laboratory evidence of infection per inclusion criteria.
  Interventions: Drug: [F-18]MHF

INTERVENTIONS:
Drug: [F-18]MHF — Following intravenous injection of 10 ± 2 mCi (370 ± 74 MBq) [F-18]MHF as a bolus, dynamic PET imaging of the lower limbs will be acquired for approximately 90 minutes. The acquired images will be processed. The uptake pattern of [F-18]MHF around infected orthopedic knee implant will be determined and compared with its uptake pattern around non-infected knee implants.
  Other Names: Fluorine-18 Maltodextrin

SUMMARY:
Following intravenous injection of [F-18]MHF as a bolus, dynamic PET imaging of the lower limbs will be acquired for approximately 90 minutes. The acquired images will be processed and viewed on a MIMVista or similar workstation. The uptake pattern of [F-18]MHF around infected orthopedic knee implant will be determined and compared with its uptake pattern around non-infected knee implants.

This study will look at how [18F]MHF goes into normal knee replacements and those with suspected infection.

DETAILED DESCRIPTION:
This is a study that will test a compound (chemical substance) that has a small amount of radioactivity attached to it. This substance has a natural tendency to go to bacterial infections. The substance is called [18F]MHF and it is given in the form of an injection into a vein. After the substance reaches the infected body region, scans called PET or Positron Emission Tomography, are done. This is similar to having CAT scans or x-rays. Usually a compound called [18]FDG is used for PET scans to detect bacterial infections but this substance can't distinguish between bacterial infections and inflammation. This substance called [18F]MHF does not go to inflamed tissue and may allow bacterial infections to be seen better.

This study will look at how [18F]MHF goes into normal knee replacements and those with suspected infection. This will hopefully lead to the development of better imaging techniques to look at bacterial infections. [18F]MHF is approved by the FDA (Food and Drug Administration) for research.

ELIGIBILITY:
Inclusion Criteria for symptomatic patient cohort

* Patients must be 18 years of age or older, able to provide written informed consent, and ability to lie still for PET scanning.
* Suspected knee prosthetic infection at least 2 months after original prosthesis placement and who are scheduled to undergo surgery debridement/removal based on the clinical assessment of the referring surgeon.
* Elevated CRP and ESR

Exclusion Criteria for symptomatic patient cohort:

* Undergoing current or recent antimicrobial therapy (within 1 month)
* Significant comorbidity such as renal failure, septic shock, uncontrolled diabetes
* Other clinically likely site of infection

Inclusion Criteria for asymptomatic cohort:

* Patients must be 18 years of age or older, able to provide written informed consent and ability to lie still for PET scanning
* Knee prosthesis in situ without complications for 6 months or longer

Exclusion Criteria for asymptomatic cohort:

* Clinical or laboratory suspicion of knee prosthesis infection
* Recent (within 3 months) or current treatment for infected knee prosthesis
* Significant comorbidity such as renal failure, septic shock, uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To accomplish the objectives of this proposed study, 20 patients symptomatic for infection of knee prosthesis and 10 patients asymptomatic for infection of knee of their prosthesis will be accrued, each receiving one injection of [F-18]MHF followed by 90 minutes dynamic PET/CT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are positive on [F-18]MHF who also have orthopedic implant-associated infections as established by the standard of truth during surgery | 2 weeks (14 days) after surgery
  Number of patients who are positive on [F-18]MHF who also have orthopedic implant-associated infections as established by the standard of truth during surgery

SECONDARY OUTCOMES:
Number of patients who are negative on [F-18]MHF who do not have have orthopedic implant-associated infections as established by the standard of truth during surgery or on clinical examination if surgery not performed. | 2 weeks (14 days) after surgery
  Number of patients who are negative on [F-18]MHF who do not have have orthopedic implant-associated infections as established by the standard of truth during surgery or on clinical examination if surgery not performed.

CONTACTS AND LOCATIONS:
Overall Officials: David Schuster, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No